CLINICAL TRIAL: NCT05720923
Title: Analysis of Muscle Morphological and Electromechanical Properties in Patients With MFS and EDS: a Low-risk Intervention Study
Brief Title: Analysis of Muscular Properties in Patients With MFS and EDS
Acronym: MUSCLE
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: University of Milan (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Unit Director, IRCCS Policlinico S. Donato
Other Study IDs: MUSCLE
Record Dates: First submitted 2023-01-19; First posted 2023-02-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Rare Diseases; Marfan Syndrome; Ehlers-Danlos Syndrome
Keywords: Rare Diseases;; Fatigue;; Muscle
MeSH Terms: conditions — Rare Diseases; Marfan Syndrome; Ehlers-Danlos Syndrome; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- MFS_f: Patients with Marfan syndrome with fatigue
  Interventions: Device: Analysis with Ergometer
- MFS_nf: Patients with Marfan syndrome without fatigue
  Interventions: Device: Analysis with Ergometer
- EDS_f: Patients with Ehlers Danlos syndrome with fatigue
  Interventions: Device: Analysis with Ergometer
- EDS_nf: Patients with Ehlers Danlos syndrome without fatigue
  Interventions: Device: Analysis with Ergometer
- Volunteers: Healthy adult volunteers without fatigue
  Interventions: Device: Analysis with Ergometer

INTERVENTIONS:
Device: Analysis with Ergometer — The analysis with the ergometer aims at assessing neuromuscular function

SUMMARY:
The goal of this observational study is to learn and assess muscle morphological and electromechanical properties in patients affected with Marfan syndrome (MFS) and Ehlers Danlos syndrome (EDS). the main questions it aims to answer are:

* To assess the ability to develop muscle strength;
* Muscle and tendon morphology involved in muscle contractions/relaxation;
* Neuromuscular functionality.

Participants will be take part in the study by performing a test for the assessment of the neuromuscular activity (voluntary muscle contractions) and undergoing a muscle ultrasound for the study of muscles and tendons.

Researchers will compare the two groups with a control group to see potential differences in the morphological and neuromuscular structures of syndromic patients.

DETAILED DESCRIPTION:
MFS, with an autosomal dominant inheritance, can lead to the presence of pathological systemic/syndromic phenotypes. Despite the cardiovascular involvement is responsible for the high mortality and morbidity, the skeletal system and the muscular system also present alterations at the metabolic level.

Like MFS, Ehlers-Danlos Syndrome (EDS) is a rare autosomal dominantly inherited connective tissue disorder. EDS is caused by mutations that cause impaired collagen production, therefore of pathological phenotypes affecting connective tissues such as the integumentary system, the system skeletal system, the cardiovascular system and other organs and tissues. Joint dislocations, musculoskeletal pain, atrophic scarring, and severe scoliosis may occur in patients with EDS.

To date, there are no studies in literature assessing neuromuscular properties in patients with MFS and EDS.

However, the analysis of the musculo-tendon morphological and mechanical properties makes it possible to evaluate the muscle capacity especially in pathological conditions, where the morphology and tendon mechanics are altered, thus providing pivotal information on changes in the contractile capacity of the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Marfan syndrome or Ehlers Danlos syndrome currently in follow-up at Cardiovascular Genetic Centre IRCCS Policlinico San Donato;
* Signed informed consent;

Exclusion Criteria:

* Previous muscle-tendon injuries in the lower and/or upper limbs;
* Presence of cardiac pacemaker;
* Epilepsia;
* Presence neurological disorders or circulatory diseases in the lower limbs;
* Pregnancy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Morphological analysis | 20 minutes
  Non invasive analysis of the tissue through ultrasound of the leg
Neuromuscular properties | 15 seconds
  Voluntary muscle contractions
Neuromuscular properties | 40 minutes
  transcutaneous electrical stimulation in electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Giuliana Trifirò, MD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy